CLINICAL TRIAL: NCT03951623
Title: The Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-523, a Syk Inhibitor in Adult Patients of Immune Thrombocytopenia: a Randomized, Double Blinded, Placebo Controlled Phase Ib Study
Brief Title: The Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-523 in Immune Thrombocytopenia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-523-00CH1
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: syk inhibitor; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Active Comparator): Eligible subjects will be treated with planned dose of 100 mg, 200 mg and 300 mg HMPL-523 once daily for 8 weeks and 16 weeks open-label treatment.
  Interventions: Drug: HMPL-523
- placebo arm (Placebo Comparator): Eligible subjects will be treated with HMPL-523 matching placebo once daily for 8 weeks and 16 weeks open-label treatment.
  Interventions: Drug: HMPL-523; Drug: Placebo

INTERVENTIONS:
Drug: HMPL-523 — HMPL-523 will be oral administrated once daily for 8 weeks and 16 weeks open-label treatment.
Drug: Placebo — HMPL-523 matching placebo will be oral administrated once daily for 8 weeks and 16 weeks open-label treatment.
  Arms: placebo arm

SUMMARY:
This is a randomized, double blinded, placebo-controlled phase Ib clinical trial in adult patients with immune thrombocytopenia. Cross-over treatment will be allowed during the study.

DETAILED DESCRIPTION:
Approximate 51 to 60 patients will be enrolled in dose escalation (3 cohorts, 8-20 subjects each with the ratio of 3:1 vs Placebo) .

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. 18~75 years old male of female
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Diagnosed immune thrombocytopenia before randomization with platelet decrease for more than 6 months.
5. Patients with refractory or relapsed ITP who have been treated with 1st line anti-ITP regimen or have experienced splenectomy.
6. Relative stable disease with World Health Organization (WHO) bleeding score of 0-1 and no rescue treatment needed within 2 weeks based on investigator's judgment.
7. Laboratory tests meet the following conditions：

   * During screening stage, twice PLT<30x10^9/L(exceed 24 hours)
   * Hb≥90g/L(if iron-deficiency anemia,Hb>80g/L),WBC>2.5x10^9/L, NEU>1.8x10^9/L
   * Crea≤1.5xULN and CCR≥50mL/min
   * TBIL、ALT、AST≤1.5xULN
   * Amylase、lipase<ULN
   * INR、APTT<20%xULN

Exclusion Criteria:

1. Patients with secondary thrombocytopenia or patients have other auto immune diseases who need long term steroids or immunosuppressants treatment.
2. Patients with Myelofibrosis, Myelodysplastic syndrome, Aplastic anemia, or other hematologic malignancies.
3. Have splenectomy within 12 weeks before randomization
4. Major surgery was performed within 4 weeks before randomization;Or require major elective surgery during the study period.
5. Have malignant tumor(except basal cell carcinoma of skin and carcinoma in situ of cervix)
6. Have previous/significant arterial/venous embolic disease
7. History of serious cardiovascular disease, or QTc≥450 ms.
8. Patients with resistant hypertension (Systolic blood pressure ≥140 mmHg or Diastolic blood pressure ≥90 mmHg)
9. Has a history of severe gastrointestinal diseases, such as dysphagia, active gastric ulcer, and is unable to take oral medication or has absorption disorder
10. HIV infection
11. Uncontrolled, active infections
12. Known history of clinically significant liver disease, such as hepatitis b（HBV DNA ≥2000IU/mL (or ≥1×104 copies)）, hepatitis c, or cirrhosis
13. Prior anti-ITP emergency treatment within 2 weeks before randomization.
14. Prior anti-ITP treatment within 4 weeks before randomization except for stable dose steroids, including but not limited to Thrombopoietin, thrombopoietin receptor agonist, azathioprine, cyclosporine A and mycophenolate mofetil.
15. Any condition requiring anti-coagulant therapy or the regular use of any medication having effluence to Platelet function.
16. Exposure to Rituximab 14 weeks prior to randomization.
17. Treament with Chinese medicine within 1 week before randomization.
18. Use of strong cytochrome P450 isoform 3A inhibitors and inducers and drugs metabolized by cytochrome P450 isoform 3A, cytochrome P450 isoform 2B6, and cytochrome P450 isoform 1A2, and are identified as narrow therapeutic drugs within 14 days or 5 half-lives, whichever is longer, prior to initiation of study treatment.
19. Prior treatment with any spleen tyrosine kinase (SYK) inhibitors (eg, fostamatinib)
20. Allergic to study drug active ingredient or excipient
21. Subjects who have participated in clinical studies of drugs or invasive medical devices within 4 week before randomization
22. Subjects have severe psychological or mental abnormalities
23. Alcoholic or drug abuser
24. Female subjects during pregnancy and lactation
25. The investigator considered that the subjects were not suitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with any Adverse Event | From first dose to within 28 days after the last dose
  Adverse Events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 15, 16, 29, 43 and 47
  Maximum plasma concentration (Cmax)
Area under the concentration-time curve in a selected time interval (AUC0-t) | Day 15, 16, 29, 43 and 47
  Area under the concentration-time curve in a selected time interval (AUC0-t)
Rate of Clinical Remission | Day 1 to 8 weeks treatment
  Rate of Clinical Remission was defined as the proportion of patients with two consecutive visits in the first 8 weeks (including the 8th week) during the medication period, platelet count ≥30×10^9/L, and a 2-fold increase from baseline (no emergency treatment during the period)

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Yin, Study Director — Hutchison Medipharma Limited
Locations (1):
- Blood diseases hospital, Chinese academy of medical university, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu X, Zhou H, Hu Y, Yin J, Li J, Chen W, Huang R, Gong Y, Luo C, Mei H, Ding B, Gu C, Sun H, Leng Y, Ji D, Li Y, Yin H, Shi H, Chen K, Wang J, Fan S, Su W, Yang R. Sovleplenib (HMPL-523), a novel Syk inhibitor, for patients with primary immune thrombocytopenia in China: a randomised, double-blind, placebo-controlled, phase 1b/2 study. Lancet Haematol. 2023 Jun;10(6):e406-e418. doi: 10.1016/S2352-3026(23)00034-0. Epub 2023 Apr 4. PMID 37028433